CLINICAL TRIAL: NCT03894553
Title: Stereotactic MRI-guided Focused Ultrasound Mesencephalotomy for Pain Palliation in Head & Neck Cancer
Brief Title: Focused Ultrasound (FUS) Mesencephalotomy for Head & Neck Cancer Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jeff Elias, MD (Other)
Responsible Party: Sponsor-Investigator, Jeff Elias, MD, Professor of Neurological Surgery, University of Virginia
Organization: University of Virginia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSR180040
Record Dates: First submitted 2018-11-12; First posted 2019-03-28 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Cancer of Head and Neck; Pain, Face; Pain, Neck
MeSH Terms: conditions — Head and Neck Neoplasms; Facial Pain; Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- FUS Mesencephalotomy (Experimental): Subjects will receive unilateral stereotactic focused ultrasound mesencephalotomy using the ExAblate Neuro device for severe, opioid-resistant pain associated with head and neck cancer.
  Interventions: Device: ExAblate Neuro

INTERVENTIONS:
Device: ExAblate Neuro — Unilateral stereotactic focused ultrasound lesioning of the contralateral mesencephalon

SUMMARY:
This proposed pilot study will investigate the safety and initial effectiveness of focused ultrasound lesioning of the contralateral mesencephalon for severe, opioid-resistant pain associated with head and neck cancer

DETAILED DESCRIPTION:
This pilot study is designed as a prospective, open-label clinical trial of stereotactic FUS mesencephalotomy in 6 subjects with treatment-refractory pain from head and neck cancer. Primary safety assessments will be made throughout the study period of 6 months following the procedure. Primary efficacy outcome is determined by comparing the difference in baseline NPRS to 3 months post treatment. All subjects receiving treatment will be followed for the six month study period.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, between 18 and 75 years, inclusive
2. Subjects with head and neck cancer, including one of the following:

   * Cancer that arises in the head and neck region: nasal cavity, sinuses, lips, mouth, salivary glands, throat, or larynx (typically squamous cell carcinoma)
   * Cancer occurring in the nasopharynx, skin, thyroid gland, and eye
   * Lymphoma
   * Sarcoma
3. Craniofacial or cervical pain related to the cancer that meets all of the following criteria:

   * Severe defined by: Worst NPRS score of ≥ 5 out of 10 at current visit and the subject reports having a similar level of pain for at least the past two months.
   * Pain is medication-refractory to all three tiers of the WHO cancer pain ladder. Thus, adequate trials of at least 3 prescription medications that will include a 'weak' and a 'strong' opioid. An adequate medication trial is defined as a therapeutic dose of each medication without sufficient effect.
   * Duration of greater than 6 months
4. Mesencephalon contralateral to the pain can be targeted by the ExAblate Neuro device. The region of the mesencephalon must be apparent on MRI. Additional MRI sequences including inversion-recovery and DTI may be utilized to refine the target.
5. Subjects who are able and willing to give consent and able to attend all study visits
6. Subjects who are able to communicate sensations during the focused ultrasound treatment

Exclusion Criteria:

1. Idiopathic trigeminal neuralgia
2. Trigeminal neuropathic pain from trauma, infection, or iatrogenic
3. Post-herpetic neuralgia
4. Headache syndromes like migraine, cluster headache
5. Temporomandibular joint syndrome
6. Atypical facial pain or pain related to a somatoform disorder
7. Subjects deemed poor candidates by a multidisciplinary team of cancer and palliative care clinicians:

   1. Significant clinician concern about reliability of subject-reported information, such as subject in active process of seeking disability for neuropathic pain
   2. Subjects exhibiting any behavior(s) consistent with ethanol or substance abuse as defined by the criteria outlined in the DSM-V as manifested by one (or more) of the following occurring within a 12 month period: Recurrent substance use resulting in a failure to fulfill major role obligations at work, school, or home (such as repeated absences or poor work performance related to substance use; substance-related absences, suspensions, or expulsions from school; or neglect of children or household). Recurrent substance use in situations in which it is physically hazardous (such as driving an automobile or operating a machine when impaired by substance use)
   3. Recurrent substance-related legal problems (such as arrests for substance related disorderly conduct)
   4. Continued substance use despite having persistent or recurrent social or interpersonal problems caused or exacerbated by the effects of the substance (for example, arguments with spouse about consequences of intoxication and physical fights).
8. Subjects with active psychiatric illness will be excluded. For the purpose of this study, active psychiatric illness includes:

   1. Exhibiting current suicide ideation and/or a history of suicide attempt within past 2 years
   2. been hospitalized for the treatment of a psychiatric illness within the past 2 years
   3. received transcranial magnetic stimulation for depression treatment
   4. received electroconvulsive therapy for depression
   5. any presence or history of psychosis
9. Subjects with unstable cardiac status including:

   1. Unstable angina pectoris on medication
   2. Subjects with documented myocardial infarction within six months of protocol entry
   3. Significant congestive heart failure defined with ejection fraction < 40
   4. Subjects with unstable ventricular arrhythmias
   5. Subjects with atrial arrhythmias that are not rate-controlled
10. Severe hypertension (diastolic BP > 100 on medication)
11. Subjects with standard contraindications for MR imaging such as non-MRI compatible implanted metallic devices including cardiac pacemakers, size limitations, etc.
12. On medications that increases the bleeding risk, based on the published guidelines which are currently recognized by the American Society of Regional Anesthesia and Pain Medicine, American Academy of Pain Medicine and the North American Neuromodulation Society (Reg Anesth Pain Med 2015;40: 182-212); specifically:

    1. Aspirin or another antiplatelet medication (clopidogrel, prasugrel, ticlopidine, abciximab) for the last 7 days prior to treatment.
    2. Oral, subcutaneous or intravenous anticoagulant medications, such as oral vitamin K inhibitors for the last 7 days, non-vitamin K inhibitor oral anticoagulant (dabigatran, apixaban, rivaroxaban) for the last 72 hours.
    3. Intravenous or subcutaneous heparin-derived compounds for the last 48 hours.
13. Individuals who are not able or willing to tolerate the required prolonged stationary supine position during treatment (can be up to 4 hours of total table time.)
14. Subjects participating or have participated in another clinical trial in the last 30 days
15. Subjects with risk factors for intraoperative or postoperative bleeding from a documented coagulopathy or if their serum coagulation studies (platelet count, PT, PTT, and INR) exceed the institutional laboratory limits.
16. Subjects with brain tumors or any significant intracranial mass.
17. Any illness that in the investigator's opinion preclude participation in this study
18. Pregnancy or lactation
19. Legal incapacity or limited legal capacity
20. Subjects with a deep brain stimulation implant
21. Skull density ratio, calculated from the baseline non-contrasted head CT, is less than 0.4
22. History of hemorrhagic stroke or cerebrovascular event within the past year of treatment exhibiting incomplete resolution
23. Subjects whose primary pain is other than craniofacial neuropathic pain.
24. Patients deemed high risk because of their airway for the procedure as evaluated by anesthesia.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 6 months post-intervention
  Number of participants with treatment-related adverse events, as assessed from adverse event reporting throughout the 6 month study period. Additional measures of safety will be made with MRI evaluation.
Numeric Pain Rating Scale | 3 months post-intervention (will also be assessed at 7 days, 1 month, and 6 months post-intervention)
  Will compare the change of WORST pain experienced in 24 hours before (baseline) and at 3 months following unilateral FUS mesencephalotomy as determined from the 11-point numeric pain rating scale (0-10), with 0 being no pain and 10 being the worst pain imaginable.

SECONDARY OUTCOMES:
Patient Global Impression of Change | Baseline, 7 days, 1 month, 3 months, and 6 months post-intervention
  Change from baseline scores to post-intervention time points (see below), as measured by a patient questionnaire that asks patients to describe the change (if any) compared to their condition prior to treatment in activity, limitations, symptoms, emotions, and overall quality of life, related to their painful condition. The options include no change, almost the same, a little better, somewhat better, moderately better, better, and a great deal better.
PROMIS scale v1.0 - Pain Intensity 3a | Baseline, 7 days, 1 month, 3 months, and 6 months post-intervention
  Change from baseline scores to post-intervention time points (see below). The first two items in the Pain Intensity item bank assess pain intensity utilizing a 7-day recall period (items include the phrase "the past 7 days") while the last item asks patient to rate their pain intensity "right now." The Pain Intensity instrument is available for adults (ages 18+). Scale includes range from 1-5, with 1 = "Had no pain" and 5 = "Very severe".
PROMIS scale v2.0 - Neuropathic Pain Quality 5a | Baseline, 7 days, 1 month, 3 months, and 6 months post-intervention
  Change from baseline scores to post-intervention time points (see below), as assessed by patient questionnaire that asks about pain quality in the past 7 days, specifically asking if the pain has felt like pins and needles, tingly, stinging, electrical, or numb, on a scale from 1-5, with 1 = "Not at all" and 5 = "Very much".
PROMIS scale v2.0 - Nociceptive Pain Quality 5a | Baseline, 7 days, 1 month, 3 months, and 6 months post-intervention
  Change from baseline scores to post-intervention time points (see below), as assessed by patient questionnaire that asks about pain quality in the past 7 days, specifically asking if the pain has felt sore, tender, achy, deep, or steady, on a scale from 1-5, with 1 = "Not at all" and 5 = "Very much".
PROMIS scale v1.0 - Pain Behavior 7a | Baseline, 7 days, 1 month, 3 months, and 6 months post-intervention
  Change from baseline scores to post-intervention time points (see below), as assessed by patient questionnaire that measures self-reported external manifestations of pain in the past 7 days, including actions and reactions that can be either verbal or nonverbal, and involuntary or deliberate. Measured on a scale from 1-6, with 1 = "Had no pain" and 6 = "Always".
PROMIS scale v1.0 - Pain Interference 8a | Baseline, 7 days, 1 month, 3 months, and 6 months post-intervention
  Change from baseline scores to post-intervention time points (see below), as assessed by patient questionnaire that measures self-reported consequences of pain on relevant aspects of one's life in the past 7 days. Includes the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities. Also incorporates items probing sleep and enjoyment in life. Measured on scale from 1-5, with 1 = "Not at all" and 5 = "Very much".
PROMIS - Ca Item Bank v1.0 - Emotional Distress-Anxiety | Baseline, 7 days, 1 month, 3 months, and 6 months post-intervention
  Change from baseline scores to post-intervention time points (see below), as assessed by patient questionnaire that measures self-reported fear (fearfulness, panic), anxious misery (worry, dread), hyperarousal (tension, nervousness, restlessness), and somatic symptoms related to arousal (racing heart, dizziness), in the past 7 days. Measured on scale from 1-5, with 1 = "Never" and 5 = "Always".
PROMIS - Ca Item Bank v1.0 - Emotional Distress-Depression | Baseline, 7 days, 1 month, 3 months, and 6 months post-intervention
  Change from baseline scores to post-intervention time points (see below), as assessed by patient questionnaire that measures self-reported negative mood (sadness, guilt), views of self (self-criticism, worthlessness), and social cognition (loneliness, interpersonal alienation), as well as decreased positive affect and engagement (loss of interest, meaning, and purpose), in the past 7 days. Somatic symptoms (changes in appetite, sleeping patterns) are not included, which eliminates consideration of these items' confounding effects when assessing patients with comorbid physical conditions. Measured on a scale from 1-5, with 1 = "Never" and 5 = "Always".
PROMIS - Ca Item Bank v1.0 - Fatigue | Baseline, 7 days, 1 month, 3 months, and 6 months post-intervention
  Change from baseline scores to post-intervention time points (see below), as assessed by patient questionnaire that measures a range of self-reported symptoms, from mild subjective feelings of tiredness to an overwhelming, debilitating, and sustained sense of exhaustion that likely decreases one's ability to execute daily activities and function normally in family or social roles. Fatigue is divided into the experience of fatigue (frequency, duration, and intensity) and the impact of fatigue on physical, mental, and social activities. The Fatigue short form is universal rather than disease-specific. It assesses fatigue over the past seven days. Measured on a scale from 1-5, with 1 = "Never" and 5 = "Always".
PROMIS - Ca Bank v1.1 - Physical Function | Baseline, 7 days, 1 month, 3 months, and 6 months post-intervention
  Change from baseline scores to post-intervention time points (see below), as assessed by patient questionnaire that measures self-reported capability rather than actual performance of physical activities. Measured on a scale from 5 to 1, with 5 = "Without any difficulty" and 1 = "Unable to do".
Pain Catastrophizing Scale | Baseline, 7 days, 1 month, 3 months, and 6 months post-intervention
  Change from baseline scores to post-intervention time points (see below), as assessed by patient questionnaire that asks participants to reflect on past painful experiences, and to indicate the degree to which they experienced each of 13 thoughts or feelings when experiencing pain, on 5-point scales with the end points (0) not at all and (4) all the time.
Daily morphine equivalents (milligrams) | Baseline, 7 days, 1 month, 3 months, and 6 months post-intervention
  Change of the amount of morphine that is used by patient daily, in daily morphine equivalents (in milligrams), from baseline through 6 months post-intervention.
Location of lesion in the x, y, z dimensions in mm | 7 days and 3 months post-intervention
  The location of the lesion will be measured in the x, y, and z dimensions, and will be reported in mm.
Precision of lesion in the x, y, z dimensions and two dimensional radial vector in mm | 7 days and 3 months post-intervention
  The precision of the lesion will be measured in the x, y, and z dimensions, but also in a two dimensional radial vector, all reported in mm.
Volume of lesion in mm3 | 7 days and 3 months post-intervention
  The volume of the lesion will be measured in mm3.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Elias, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia UVA Health, University Hospital, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No